CLINICAL TRIAL: NCT03179813
Title: Topical Hydrocortisone for Pain and Edema Control After Third Molar Surgery: a Clinical, Crossover, Randomized, Double-blind, Controlled Study
Brief Title: Topical Hydrocortisone for Pain and Edema Control After Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Vitor Pereira Rodrigues, PhD candidate, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 44657315.4.0000.0075
Record Dates: First submitted 2017-05-29; First posted 2017-06-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2017-11

CONDITIONS: Impacted Third Molar Tooth
Keywords: hydrocortisone; third molar; oral surgery; postoperative pain; edema
MeSH Terms: conditions — Pain, Postoperative; Edema | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone group (Experimental): Intraoperative topical use of hydrocortisone as a irrigation solution in third molar surgery.
  Interventions: Procedure: Hydrocortisone
- Control Group (Placebo Comparator): Intraoperative irrigation with saline solution.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Hydrocortisone — During the third molar extraction the hydrocortisone solution will be used in the test group
  Arms: Hydrocortisone group
Procedure: Control — During the third molar extraction the saline solution will be used in the control group
  Arms: Control Group

SUMMARY:
The investigators set out to develop a clinical trial in order to test the topical use of hydrocortisone as a intraoperative irrigant solution. As this route of administration as well as being low cost and not add new steps to the surgical procedure, can contribute to an improved quality of life in the postoperative period of patients undergoing extraction of third molars.

DETAILED DESCRIPTION:
Third molars are the teeth with a higher prevalence of failure in eruption and surgery for extraction of these impacted teeth is one of the most commonly procedures performed by the oral and maxillofacial surgeon. In most cases these are not traumatic procedures, however factors such as patient age, habits, degree of tooth impaction and surgeon experience can influence the surgical trauma and therefore the postoperative period could include swelling and pain of varying magnitudes which can significantly affect the patient's quality of life.

The study is designed as a prospective, randomized, placebo-controlled, split-mouth crossover trial. All the patients will be informed of the experimental methodology and signed a institutionally approved consent form. The study is been conducted in compliance with Declaration of Helsinki (1989), and was revised by the Institutional Ethical Committee (protocol 1.167.908).

ELIGIBILITY:
Inclusion Criteria:

* Health patients of any sex, with symmetric bilateral bone-impacted mandibular third molars requiring surgical removal, and with no history of allergy to the drugs used in this study.

Exclusion Criteria:

* Use of analgesic or anti-inflammatory drugs 24 hours before the surgery.
* Pregnant or breastfeeding patients,
* Use of other drugs beyond of that one's prescribed by the researchers;

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Edema | From the preoperative moment to the second postoperative day
  Change in edema measures

SECONDARY OUTCOMES:
Pain | Up to 2 days (amount of analgesic medication intake form the immediate postoperative moment to the second postoperative day)
  Quantitative evaluation (amount of analgesic medication intake)
Pain | Up to 2 days (from the immediate postoperative moment to the second postoperative day)
  Subjective evaluation - Visual Analog Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Vitor Pereira Rodrigues, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngeow WC, Lim D. Do Corticosteroids Still Have a Role in the Management of Third Molar Surgery? Adv Ther. 2016 Jul;33(7):1105-39. doi: 10.1007/s12325-016-0357-y. Epub 2016 Jun 10. PMID 27287853
- [Background] Herrera-Briones FJ, Prados Sanchez E, Reyes Botella C, Vallecillo Capilla M. Update on the use of corticosteroids in third molar surgery: systematic review of the literature. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 Nov;116(5):e342-51. doi: 10.1016/j.oooo.2012.02.027. Epub 2012 Aug 17. PMID 22902498
- [Background] Grossi GB, Maiorana C, Garramone RA, Borgonovo A, Beretta M, Farronato D, Santoro F. Effect of submucosal injection of dexamethasone on postoperative discomfort after third molar surgery: a prospective study. J Oral Maxillofac Surg. 2007 Nov;65(11):2218-26. doi: 10.1016/j.joms.2006.11.036. PMID 17954317
- [Background] Ceccheti MM, Negrato GV, Peres MP, Deboni MC, Naclerio-Homem Mda G. Analgesic and adjuvant anesthetic effect of submucosal tramadol after mandibular third molar surgery. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Mar;117(3):e249-54. doi: 10.1016/j.oooo.2012.05.015. Epub 2012 Sep 12. PMID 22981094
- [Background] Pourdanesh F, Khayampour A, Jamilian A. Therapeutic effects of local application of dexamethasone during bilateral sagittal split ramus osteotomy surgery. J Oral Maxillofac Surg. 2014 Jul;72(7):1391-4. doi: 10.1016/j.joms.2013.12.025. Epub 2014 Jan 15. PMID 24576440
- [Background] Mahmoud Hashemi H, Mohammadi F, Hasheminasab M, Mahmoud Hashemi A, Zahraei S, Mahmoud Hashemi T. Effect of low-concentration povidone iodine on postoperative complications after third molar surgery: a pilot split-mouth study. J Oral Maxillofac Surg. 2015 Jan;73(1):18-21. doi: 10.1016/j.joms.2014.06.454. Epub 2014 Jul 5. PMID 25249172
- [Background] UStun Y, Erdogan O, Esen E, Karsli ED. Comparison of the effects of 2 doses of methylprednisolone on pain, swelling, and trismus after third molar surgery. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Nov;96(5):535-9. doi: 10.1016/S1079210403004645. PMID 14600686